CLINICAL TRIAL: NCT02104830
Title: Multicenter Randomized Double-blind Phase III Clinical Study Comparing the Efficacy and Safety of a Single Dose Extimia® Versus Daily Filgrastim for Neutropenia Prophylaxis in Breast Cancer Patients Receiving Myelosuppressive Chemotherapy
Brief Title: Study of the Efficacy and Safety of Empegfilgrastim for Neutropenia Prophylaxis in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BCD-017-3
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: empegfilgrastim; pegylated filgrastim; neutropenia; febrile neutropenia; chemotherapy-associated neutropenia; breast cancer; docetaxel; doxorubicin
MeSH Terms: conditions — Neutropenia; Febrile Neutropenia; Breast Neoplasms | interventions — Filgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Empegfilgrastim 6 mg (Experimental): Patients will receive a single administration of empegfilgrastim at a dose of 6 mg subcutaneously, 24 h after the chemotherapy and placebo #2 in a dose of 0.0083 ml/kg in 24-27 hour after chemotherapy, then patient received placebo #2 in dose 0.0083 ml/kg until ANC ≥ 10x109/L or during 14 days
  Interventions: Biological: Empegfilrastim 6 mg; Biological: Placebo №2
- Empegfilgrastim 7.5 mg (Experimental): Patients will receive a single administration of empegfilgrastim at a dose of 7.5 mg subcutaneously, 24 h after the chemotherapy and placebo #2 in a dose of 0.0083 ml/kg in 24-27 hour after chemotherapy, then patient received placebo #2 in dose 0.0083 ml/kg until ANC ≥ 10x109/L or during 14 days
  Interventions: Biological: Placebo №2; Biological: Empegfilrastim 7.5 mg
- Filgrastim (Active Comparator): Patients will receive filgrastim at a dose of 5 μg/kg subcutaneously daily (until ANC 10 000/μL or for 14 days, whichever occurred first), starting 24 h after the chemotherapy and placebo #1 in dose 1.0 ml subcutaneously, 24 h after the chemotherapy.
  Interventions: Biological: Filgrastim; Biological: Placebo №1

INTERVENTIONS:
Biological: Empegfilrastim 6 mg — Empegfilgrastim is supplied as solution for injection 3 mg/ml. Empegfilgrastim is to be administered 24 h after the chemotherapy at dose of 6 mg.
  Other Names: Extimia; metpegfilgrastim; pegylated filgrastim; peg-GCSF
  Arms: Empegfilgrastim 6 mg
Biological: Filgrastim — Filgrastim should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Filgrastim should be administered daily for up to 2 weeks until the ANC has reached 10 000/mm3 following the expected chemotherapy-induced neutrophil nadir.
  Other Names: GCSF
  Arms: Filgrastim
Biological: Placebo №1 — Placebo №1 is supplied as solution for injection 1.0 ml. Placebo №1 is to be administered 24 h after the chemotherapy at dose of 1.0.
  Arms: Filgrastim
Biological: Placebo №2 — Placebo №2 should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Placebo №2 is supplied as solution for injection 0.0083 ml/kg.
  Arms: Empegfilgrastim 6 mg; Empegfilgrastim 7.5 mg
Biological: Empegfilrastim 7.5 mg — Empegfilgrastim is supplied as solution for injection 3 mg/ml. Empegfilgrastim is to be administered 24 h after the chemotherapy at dose of 6 mg.
  Other Names: Extimia; metpegfilgrastim; pegylated filgrastim; peg-GCSF
  Arms: Empegfilgrastim 7.5 mg

SUMMARY:
The purpose of the study is to compare safety and efficacy of a single dose of empegfilgrastim and daily dosing of filgrastim for prevention of neutropenia in patients receiving AT (docetaxel 75 mg/m2 + doxorubicin 50 mg/m2).

DETAILED DESCRIPTION:
BCD-017-3 is an double-blind randomized phase III clinical study to compare the incidence of CTCAE grade 3/4 neutropenia after a single administration of recombinant human pegylated filgrastim empegfilgrastim (Extimia®) at a dose of 6 or 7.5 mg versus daily administration of filgrastim at a dose of 5 μg/kg/day for neutropenia prophylaxis in breast cancer patients receiving myelosuppressive chemotherapy.

The study also includes the following determination of pharmacokinetic parameters after repeated administration of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Histologically verified diagnosis of stage IIb/III/IV breast cancer;
* Age of 18-70 years inclusive;
* Life expectancy of at least 6 months after inclusion in the study;
* If the patient had received the chemotherapy for breast cancer, it should be finished 30 days before the beginning of the study;
* ECOG Performance Status of 0- 2, not increasing within during 2 weeks before randomization;
* ANC level of 1500/μL and more at the beginning of the study
* Platelet count of 100 000/μL and more at the beginning of the study
* Hemoglobin level of 90 g/l and more
* Creatinine level <1.5 mg/dl
* Total bilirubin level <1.5 × the upper limit of normal (ULN)
* ALT and/or AST levels <2.5×ULN (5×ULN for patients with liver metastases);
* Alkaline phosphatase <5×ULN;
* Left ventricular ejection fraction >50% and more;
* If the patient had received adjuvant and/or neoadjuvant therapy, the cumulative dose of anthracyclines should not exceed 250 mg/m2 for doxorubicin or 540 mg/m2 for epirubicin,if in this study planned 6 cycles of chemotherapy ;
* If the patient had received adjuvant and/or neoadjuvant therapy, the cumulative dose of anthracyclines should not exceed 350 mg/m2 for doxorubicin or 660 mg/m2 for epirubicin,if in this study planned 4 cycles of chemotherapy ;
* Ability of the participant to follow the protocol requirements, according to the Investigator's opinion;
* Patients of childbearing potential must implement reliable contraceptive measures during the study treatment, starting 4 weeks prior randomization and for 6 months after the last administration of the study drug;
* Patients should be able to follow the Protocol procedures (according to Investigator's assessment.

Exclusion Criteria:

* Patient has received two or more chemotherapy regimens for the metastatic breast cancer;
* Documented hypersensitivity to filgrastim, pegfilgrastim, docetaxel, doxorubicin, dexamethasone and/or its excipients, PEGylated drugs, recombinant proteins.
* Pregnancy or breastfeeding;
* Systemic antibiotic therapy within 72 h prior empegfilgrastim/filgrastim administration;
* Concomitant radiotherapy (except selective radiotherapy of bone metastases);
* Surgery, radiotherapy (except selective radiotherapy of bone metastases), administration of any experimental drugs within 30 days prior randomization;
* History of bone marrow/stem cell transplantation;
* Conditions limiting the patient's ability to follow the protocol;
* CTCAE grade 3-4 neuropathy;
* HIV, HCV, HBV, T.Pallidum infection(s);
* Acute or active chronic infections;
* Severe concurrent diseases (for example, severe arterial hypertension, severe heart failure, and other);
* Severe depression, schizophrenia, any other mental disorders;
* Obstacles in intravenous administration of study drugs;
* Simultaneous participation in other clinical trials, previous participation in other clinical trials within 30 days before entering into the trial, previous participation in the same trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, MD, PhD, Study Director — Biocad; Larisa Bolotina, MD, PhD, Principal Investigator — Federal State Institution "Moscow Research Oncological Institute P.A.Gertsena "of the Ministry of Health of the Russian Federation; Olga Brichkova, MD, PhD, Principal Investigator — State public health institution "Regional Oncology Dispensary №1; Olga Burdaeva, MD, Principal Investigator — State Budget Institution of Health Arkhangelsk region "Arkhangelsk Clinical Oncology Dispensary"; Byakhov Michael, MD, PhD, Principal Investigator — Non-governmental healthcare institution "Central Clinical Hospital № 2 Semashko" JSC "Russian Railways"; Vladimir Vladimirov, MD, PhD, Principal Investigator — State Budget Institution of Health Stavropol area "Piatigorsky Oncology Dispensary"; Rinat Galiulin, MD, Principal Investigator — State budget healthcare institution Omsk region "Clinical Oncology Dispensary"; Oleg Gladkov, MD, PhD, Principal Investigator — State Budget Institution of Health "Chelyabinsk Regional Clinical Oncology Dispensary"; Irina Davydenko, PhD, Principal Investigator — State Budget Institution of Health "Clinical Oncology Dispensary № 1" of the Ministry of Health of the Krasnodar area; Victoria Elkova, MD, Principal Investigator — State public health institution "Voronezh Regional Clinical Oncology Dispensary"; Igor Lifirenko, MD, Principal Investigator — State public health institution "Kursk Regional Oncology Dispensary"; Nadezhda Kovalenko, PhD, Principal Investigator — State Budget Institution of Health "Volgograd regional oncologic dispensary № 3"; Michael Kopp, MD, PhD, Principal Investigator — State Budget Institution of Health "Samara Regional Clinical Oncology Dispensary"; Bogdan Kotiv, MD, PhD, Principal Investigator — S. M. Kirov Military Medical Academy of the Ministry of Defense of the Russian Federation; Natalia Levchenko, PhD, Principal Investigator — State Budget Institution of Health Stavropol area "Stavropol Regional Clinical Oncology Dispensary"; Marina Matrosova, MD, Principal Investigator — State public health institution "Nizhny Novgorod Regional Oncology Dispensary"; Guzel Mukhametshina, MD, Principal Investigator — State public health institution "Republican Clinical Oncology Dispensary" of the Ministry of Health of the Republic of Tatarstan; Sergei Panchenko, PhD, Principal Investigator — State public health institution "Regional Clinical Oncology Dispensary"; Alexander Pecheny, PhD, Principal Investigator — Regional State Health Care Institution "Orlovsky Oncology Dispensary"; Igor Pimenov, PhD, Principal Investigator — State Budget Institution health care "Tula Regional Oncology Dispensary"; Andrei Sinykov, PhD, Principal Investigator — State Health Care Institution of Tyumen Region "Regional Oncological Dispensary"; Pavel Skopin, PhD, Principal Investigator — Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva "; Daniil Stroyakovsky, Principal Investigator — State Health Care Institution "Moscow City Oncology Hospital № 62" Moscow Health Department; Sergei Tyulyandin, MD, PhD, Principal Investigator — "Russian Oncological Scientific Center N.N.Blokhin" Russian Academy of Sciences; Dmitriy Udovica, MD, Principal Investigator — State Health Care Institution "Oncologic Dispensary № 2" Health Department of Krasnodar Area; Andrei Horinko, MD, Principal Investigator — State Health Care Institution "Perm Regional Oncology Dispensary"; Petr Krivorotko, MD, Principal Investigator — N.N. Petrov Oncology Research Center of the Ministry of Health of the Russian Federation; Yulia Shapovalova, PhD, Principal Investigator — Non-governmental healthcare institution "Chelyabinsk Road Clinical Hospital" JSC "Russian Railways"; Ludmila Sheveleva, MD, Principal Investigator — State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1"; Vadim Shirinkin, MD, Principal Investigator — State Health Care Institution "Orenburg Regional Clinical Oncology Dispensary"; Shekar Patil, MD, Principal Investigator — Bangalore Institute of Oncology; Prasad Narayanan, MD, Principal Investigator — Mazumdar Shaw Cancer Center and Narayana Hrudayalaya Multispecialty Hosptial; Nalini Kilara, MD, Principal Investigator — M.S.Ramaiah Memorial Hospital; Sergei Kulik, MD, Principal Investigator — Donetsk City Municipal Oncology Dispensary; Igor Sedakov, MD, PhD, Principal Investigator — Donetsk Regional oncology centers; Andrei Rusin, MD,PhD, Principal Investigator — Zakarpatskii Regional Clinical Oncology Dispensary; Yuri Vinnik, MD, PhD, Principal Investigator — Kharkiv Regional Clinical Oncology Center; Sergei Odarchenko, PhD, Principal Investigator — Vinnitskii Regional Oncology Dispensary
Locations (13):
- Russia (13):
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - Clinical Hospital at Chelyabinsk Railway Station, Chelyabinsk
  - State public health institution "Republican Clinical Oncology Dispensary" of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - Non-governmental healthcare institution "Central Clinical Hospital № 2 Semashko" JSC "Russian Railways", Moscow
  - State Health Care Institution "Moscow City Oncology Hospital № 62" Moscow Health Department, Moscow
  - State public health institution "Nizhny Novgorod Regional Oncology Dispensary", Nizhny Novgorod
  - Perm Region Oncology Dispensary, Perm
  - Pyatigorsk Oncology Center, Pyatigorsk
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - State public health institution "Regional Clinical Oncology Dispensary", Ulyanovsk
  - Volgograd Regional Oncology Dispensary №3, Volgograd
  - State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1", Volgograd

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patients were withdrawn for various reasons without receiving any dose of any of the studied products.
Groups:
- Empegfilgrastim 6 mg: Patients will receive a single administration of empegfilgrastim at a dose of 6 mg subcutaneously , 24 h after the chemotherapy
  Placebo №2: Placebo №2 should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Placebo №2 is supplied as solution for injection 0.0083 ml/kg.
- Empegfilgrastim 7.5 mg: Patients will receive a single administration of empegfilgrastim at a dose of 7.5 mg subcutaneously, 24 h after the chemotherapy
  Placebo №2: Placebo №2 should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Placebo №2 is supplied as solution for injection 0.0083 ml/kg.
- Filgrastim: Patients will receive filgrastim at a dose of 5 μg/kg subcutaneously daily (until ANC 10 000/μL or for 14 days, whichever occurred first), starting 24 h after the chemotherapy
  Placebo №1: Placebo №1 is supplied as solution for injection 1.0 ml. Placebo №1 is to be administered 24 h after the chemotherapy at dose of 1.0.
Period: Overall Study
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Started | 42 | 43 | 43
Completed | 38 | 36 | 36
Not Completed | 4 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Empegfilgrastim 7.5 mg: Patients will receive a single administration of empegfilgrastim at a dose of 7.5 mg subcutaneously, 24 h after the chemotherapy and placebo #2 in a dose of 0.0083 ml/kg in 24-27 hour after chemotherapy, then patient received placebo #2 in dose 0.0083 ml/kg until ANC ≥ 10x109/L or during 14 days
  Placebo №2: Placebo №2 should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Placebo №2 is supplied as solution for injection 0.0083 ml/kg.
  empegfilrastim 7.5 mg: Empegfilgrastim is supplied as solution for injection 3 mg/ml.
  Empegfilgrastim is to be administered 24 h after the chemotherapy at dose of 6 mg.
- Filgrastim: Patients will receive filgrastim at a dose of 5 μg/kg subcutaneously daily (until ANC 10 000/μL or for 14 days, whichever occurred first), starting 24 h after the chemotherapy and placebo #1 in dose 1.0 ml ubcutaneously, 24 h after the chemotherapy.
  filgrastim: Filgrastim should be administered no earlier than 24 hours after the administration of cytotoxic chemotherapy. Filgrastim should be administered daily for up to 2 weeks until the ANC has reached 10 000/mm3 following the expected chemotherapy-induced neutrophil nadir.
  Placebo №1: Placebo №1 is supplied as solution for injection 1.0 ml. Placebo №1 is to be administered 24 h after the chemotherapy at dose of 1.0.
- Total: Total of all reporting groups
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim | Total
Number analyzed (Participants) | 42 | 43 | 43 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 43 | 43 | 128
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.38 (11.07) | 50.42 (9.19) | 51.86 (9.68) | 50.23 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 43 | 128
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 42 | 43 | 43 | 128
Histologic type [Number; unit: participants]
  Infiltrative ductal | 27 | 28 | 33 | 88
  Infiltrative lobular | 6 | 3 | 2 | 11
  Medullar | 0 | 1 | 0 | 1
  Squamous cell cancer | 0 | 1 | 0 | 1
  Infiltrative not specified | 4 | 5 | 4 | 13
  Low-grade differentiated carcinoma | 2 | 3 | 1 | 6
  Undifferentiated cancer | 3 | 2 | 3 | 8
Disease stage [Number; unit: participants]
  IIA | 13 | 12 | 10 | 35
  IIB | 5 | 7 | 9 | 21
  IIIA | 5 | 7 | 10 | 22
  IIIB | 12 | 10 | 8 | 30
  IIIС | 2 | 1 | 0 | 3
  IV | 5 | 6 | 6 | 17
History previous therapy of breast cancer [Number; unit: participants] — Patients with previous therapy could be treated with several different types of therapy (for example surgery treatment and adjuvant chemotherapy)
  participants
    Adjuvant chemotherapy | 7 | 8 | 10 | 25
    Neoadjuvant chemotherapy | 1 | 1 | 0 | 2
    Radiotherapy | 8 | 4 | 3 | 15
    Hormone therapy | 6 | 7 | 4 | 17
    Surgery treatment | 28 | 27 | 22 | 77
    Any treatment | 28 | 29 | 26 | 83
Duration of a disease [Mean (Full Range); unit: months] | 16.14 [1.0 to 144.0] | 11.62 [1.0 to 144.0] | 5.37 [1.0 to 51.0] | 11.0 [1.0 to 144.0]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Neutropenia CTCAE Grade 4
Description: The primary endpoint, which will allow to compare the efficacy of the single dose of Extimia® versus nonpegylated daily filgrastim is the number of breast cancer patients developing CTCAE grade 3/4 neutropenia after the first AT chemotherapy cycle (doxorubicin+docetaxel).
Time Frame: 3 weeks
Population: The efficacy analysis included only those patients who received at least one dose of study drug, and who were participated in the study for 2 weeks or more.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
days | 0.905 (1.206) | 0.791 (1.013) | 1.725 (1.519)

2. Secondary Outcome: The Duration of Grade 4 Neutropenia From the 2nd (Week 6) to 4th Cycle (Week 12);
Time Frame: 2nd cycle (week 6), 3rd cycle (week 9), 4th cycle (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
days
  2nd cycle (week 6) | 0.452 (1.194) | 0.326 (0.919) | 0.925 (1.385)
  3rd cycle (week 9) | 0.244 (0.734) | 0.310 (0.680) | 0.641 (0.932)
  4th cycle (week 12) | 0.195 (0.601) | 0.475 (1.320) | 0.892 (1.197)

3. Secondary Outcome: The Incidence of Severe Neutropenia (Grade 3-4)
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
participants | 40 | 34 | 40

4. Secondary Outcome: Low Level (Nadir) ANC x 10^9/L
Time Frame: 1st cycle (week 3), 2nd cycle (week 6), 3rd cycle (week 9), 4th cycle (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
cells x 10^9/L
  1st cycle (week 3) | 0.68 (0.68) | 0.91 (1.11) | 0.47 (0.74)
  2nd cycle (week 6) | 1.44 (1.30) | 2.10 (1.78) | 0.87 (1.12)
  3rd cycle (week 9) | 1.77 (1.39) | 1.88 (1.71) | 0.94 (1.04)
  4th cycle (week 12) | 1.67 (1.12) | 2.07 (1.75) | 0.75 (0.87)

5. Secondary Outcome: Neutropenia Duration, Any Grade
Time Frame: 1st cycle (week 3), 2nd cycle (week 6), 3rd cycle (week 9), 4th cycle (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
days
  1st cycle (week 3) | 2.214 (1.152) | 1.953 (1.194) | 4.0 (3.121)
  2nd cycle (week 6) | 1.881 (2.276) | 1.233 (1.702) | 2.775 (2.434)
  3rd cycle (week 9) | 1.585 (1.897) | 1.024 (1.199) | 2.487 (2.480)
  4th cycle (week 12) | 1.146 (1.195) | 1.525 (2.364) | 2.919 (2.488)

6. Secondary Outcome: Duration From ANC Nadir to ANC < 2.0 x 10^9/L
Time Frame: 1st cycle (week 3), 2nd cycle (week 6), 3rd cycle (week 9), 4th cycle (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Number analyzed (Participants) | 42 | 43 | 40
days
  1st cycle (week 3) | 1.74 (0.98) | 1.51 (0.86) | 2.98 (2.40)
  2nd cycle (week 6) | 1.43 (1.29) | 1.05 (1.31) | 2.05 (1.08)
  3rd cycle (week 9) | 1.20 (1.21) | 0.98 (0.90) | 1.90 (1.87)
  4th cycle (week 12) | 1.12 (1.05) | 1.03 (1.20) | 2.14 (1.70)

ADVERSE EVENTS:
Time Frame: 3 month
Description: In general, any AEs were reported in all patients in both groups over a period of study. The vast majority of AEs were due to myelosuppressive chemotherapy. When comparing the frequency of registration of individual AEs there was no significant difference. AEs specific for all G-CSF drugs were observed rarely.
Arm/Group | Empegfilgrastim 6 mg | Empegfilgrastim 7.5 mg | Filgrastim
Serious Adverse Events (participants affected / at risk) | 1/42 | 1/43 | 5/43
Other Adverse Events (participants affected / at risk) | 42/42 | 43/43 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empegfilgrastim 6 mg (N=42) | Empegfilgrastim 7.5 mg (N=43) | Filgrastim (N=43)
Uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Left hand fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
nose furunculus 3 grade (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Empegfilgrastim 6 mg (N=42) | Empegfilgrastim 7.5 mg (N=43) | Filgrastim (N=43)
neutropenia any grade (Blood and lymphatic system disorders) | 41 (41) | 37 (37) | 41 (41)
Anemia (Blood and lymphatic system disorders) | 17 (17) | 13 (13) | 19 (19)
Leucopenia (Blood and lymphatic system disorders) | 41 (41) | 38 (38) | 41 (41)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2)
Hyperglycemia (Endocrine disorders) | 6 (6) | 8 (8) | 9 (9)
Hyperbilirubinemia (Hepatobiliary disorders) | 7 (7) | 7 (7) | 2 (2)
Liver enzymes (ALT) elevation (Hepatobiliary disorders) | 4 (4) | 2 (2) | 2 (2)
Hyperemia after injection (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Weakness / asthenia (General disorders) | 26 (26) | 24 (24) | 24 (24)
Fever (General disorders) | 2 (2) | 3 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 3 (3)
Headache (General disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes